CLINICAL TRIAL: NCT04268953
Title: A Phase 1, Single-centre, Multiple-dose, Open-label Study to Assess the Safety, Tolerability, and Pharmacokinetics of the AC-SD-03 Formulation of Tricaprilin in Healthy Older Volunteers
Brief Title: Study to Compare the Pharmacokinetics of Daily Administration of Tricaprilin on Ketone Body Production
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AC-20-021
Record Dates: First submitted 2020-02-12; First posted 2020-02-13 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tricaprylin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AC-SD-03 (Experimental): Study drug administered concurrently with a standard meal
  Interventions: Drug: Tricaprilin

INTERVENTIONS:
Drug: Tricaprilin — Tricaprilin formulated as AC-SD-03 mixed in 300mL water

SUMMARY:
This is a Phase I, single center, open label, multiple dose, pharmacokinetic (PK) study recruiting healthy older subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, males or females, age 50 years and above, at Screening.
2. Subject must be in reasonably good health as determined by the investigator based on a detailed medical history, full physical examination (including blood pressure and pulse rate measurement), 12 lead ECG and clinical laboratory tests. Subjects with mild, chronic, stable disease (e.g., controlled hypertension, Type 2 diabetes, etc) will be permitted to enrol.
3. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at Screening.
4. Agrees to comply with study procedures including the confinement period of 28 days.
5. Subject is able and willing to consume a prescribed full breakfast, lunch and dinner while confined in the CRU. Subject does not have specific dietary requirements (vegetarian, vegan, lactose-free, low-fat, etc.).
6. Subject is not consuming a ketogenic diet (defined by consumption of < 50 gm carbohydrates per day).
7. A non vasectomized male subject must agree to use a condom or abstain from sexual intercourse during the study and for 90 days following last dose of AC-SD 03. No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to Screening. A subject who has been vasectomized less than 4 months prior to Screening must follow the same restrictions as a non vasectomized male.
8. Female subjects must be either surgically sterile or 2 or more years post-menopause.
9. Has given voluntary, written informed consent to participate in the study.

Exclusion Criteria:

1. History or presence of alcoholism or substance abuse disorder within the last year.
2. Positive urine drug screen at Screening or Check-In.
3. Subject is currently actively using MCTs, ketone esters, or other ketogenic products or is following a ketogenic diet.
4. Clinically significant abnormal laboratory results at Screening that in the opinion of the PI preclude participating in this study
5. Participation in another clinical trial within 30 days prior to Check-In.
6. Subject has a known allergy to the study drug's active or inactive ingredients.
7. Subject has been following a ketogenic diet (or other diet incompatible with the on-study diet), in the opinion of the investigator.
8. Unable to refrain from, or anticipates the use of drugs other than allowed products, including prescription and non-prescription medications, beginning 14 days prior to the first dose and throughout the study.

   1. Allowed medications include anti-hypertensive agents, statins, aspirin in a dose of 100 mg or less per day for prophylaxis.
   2. Paracetamol (acetaminophen), up to 4 g per 24 hour period, or ibuprofen (up to 1200 mg per 24-hour period) may be permitted during the study.
   3. Herbal remedies and vitamin supplements are permitted in usual doses (not hyper supplementation) so long as subject has been on stable amounts for at least 6 weeks.
   4. Agents being taken to improve memory or cognition are not allowed, whether herbal, 'natural' or pharmaceutical.
9. Subject is known HIV, HBV or HCV positive, or has a positive test at Screening.
10. Any other condition which, in the investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple-dose administrations of tricaprilin formulated as AC-SD-03 administered using a titration scheme in healthy older volunteers | 32 days
  TEAE incidence rate

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameters of Total Ketones levels after multiple dose of AC-SD-03 using AUC(0-t) | 28 days
  AUC(0-t) will be calculated from PK concentrations of Total Ketones (B-hydroxybutyrate and Acetoacetate) Levels. AUC (0-t) = Area under the concentration-time curve from 0 to last quantifiable concentration. Summary statistics will be generated for each PK parameter.
Pharmacokinetics (PK) parameters of Total Ketones levels after multiple dose of AC-SD-03 using Cmax | 28 days
  Cmax will be calculated from PK concentrations of Total Ketones (B-hydroxybutyrate and Acetoacetate) Levels. Cmax = Cmax is maximum concentration, determined directly from individual concentration-time data.Summary statistics will be generated for each PK parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No